CLINICAL TRIAL: NCT05489302
Title: Evaluation of Two Protocol of Maxillary Protraction in Class III Adolescent After Using (MSE) Alt-RAMEC vs Conventional Rapid Palatal Expansion Randomized Controlled Trial -CBCT Study
Brief Title: Evaluation of Two Protocol of Maxillary Protraction in Class III Adolescent After Using (MSE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelrhman Shendy Abdelrhman, lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 828/220
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Maxillary Protraction in Class III Adolescent After Using (MSE)
Keywords: Expansion; maxillary protraction; class III

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (MSE) Alt-RAMEC protocol (Active Comparator)
  Interventions: Device: Maxillary skeletal expander with protraction face mask with Alt-RAMEC protocol.
- (MSE) conventional protocol (Active Comparator)
  Interventions: Device: Maxillary skeletal expander with protraction face mask with conventional protocol

INTERVENTIONS:
Device: Maxillary skeletal expander with protraction face mask with Alt-RAMEC protocol. — The current study was conducted on a total sample of 21 young adult orthodontic patients presented with class 3 retrognathic maxilla with or without transverse maxillary deficiency by Alt-RAMEC protocol.
  Arms: (MSE) Alt-RAMEC protocol
Device: Maxillary skeletal expander with protraction face mask with conventional protocol — The current study was conducted on a total sample of 21 young adult orthodontic patients presented with class 3 retrognathic maxilla with or without transverse maxillary deficiency by conventional protocol
  Arms: (MSE) conventional protocol

SUMMARY:
The aim of this study of this study is to compare two protocol of maxillary protraction in class III adolescent after using (MSE) Alt-RAMEC vs conventional rapid palatal expansion using cone beam computed tomography (CBCT)

ELIGIBILITY:
Inclusion Criteria:

* Class3 Patients suffering maxillary collapse with a skeletal background
* Patients with retrognathic maxilla.
* Patients with anterior cross-bite or incisor end-to-end relationship
* Patients with unilateral or bilateral posterior crossbite.
* Patients with no periodontal disease.
* Patients with good oral hygiene and general health.
* No systemic diseases that may affect bone quality or interfere with orthodontic treatment.
* Patients with no previous orthodontic treatment.

Exclusion Criteria:

* previous orthodontic treatment.
* Craniofacial syndrome.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
amount of maxillary protraction | 6 months
  protraction of maxilla using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Shendy, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No
Evaluation of two protocol of maxillary protraction in class III adolescent after using (MSE) Alt-RAMEC vs conventional rapid palatal expansion

REFERENCES:
- [Background] Liou EJ, Tsai WC. A new protocol for maxillary protraction in cleft patients: repetitive weekly protocol of alternate rapid maxillary expansions and constrictions. Cleft Palate Craniofac J. 2005 Mar;42(2):121-7. doi: 10.1597/03-107.1. PMID 15748102